CLINICAL TRIAL: NCT00326768
Title: An Open-Label, Long-term (52-week), Safety Trial of the Fixed Dose Combination of Telmisartan 80mg Plus Hydrochlorothiazide 12.5mg and Telmisartan 40mg Plus Hydrochlorothiazide 12.5mg in Patients With Essential Hypertension - Efficacy and Safety Evaluation
Brief Title: Trial of Telmisartan 80 mg/HCTZ 12.5 mg and Telmisartan 40 mg/HCTZ 12.5 mg in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.516
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan 40 mg/HCTZ 12.5 mg
Drug: Telmisartan 40 mg
Drug: Telmisartan 80 mg/HCTZ 12.5 mg

SUMMARY:
The objective of this trial is to assess the safety and efficacy of 52 weeks of open-label treatment with the fixed dose combination of telmisartan 80 mg plus HCTZ 12.5 mg and telmisartan 40 mg plus HCTZ 12.5 mg in patients with essential hypertension.

DETAILED DESCRIPTION:
This is a multi-centre study with three centres participating with a target of 30 to 90 patients entering the maintenance period and 20-60 patients completing long-term treatment per centre. The recruitment period will be about three months from the start of the study.

Study Hypothesis:

The primary objective of this study is to demonstrate the long-term safety of a fixed dose combination of telmisartan/HCTZ fixed-dose combination treatment. This study has no control group; therefore, no hypothesis testing will be performed.

Comparison(s):

This study has no control group.

ELIGIBILITY:
1. Essential hypertensive patients who meet the following criteria:

   * In case of using any antihypertensives, mean seated DBP* must be over 90 and under 114 mmHg at Visit 1
   * In case of not using any antihypertensives, mean seated DBP* must be over 95 and under 114 mmHg at Visit 1
   * Mean seated DBP* must be over 90 at Visit 2 (* The mean DBP values will be calculated as the average of three seated measurements taken at two-minute intervals).
2. Age over 20 and under 80 years at Visit 1 (Male or Female)
3. Outpatient
4. Patients who are able to stop current anti-hypertensive therapy at Visit 1 if taking any anti-hypertensive medications
5. Patients with an ability to provide written informed consent in accordance with the related laws and guidelines such as Good Clinical Practice (GCP) and the Pharmaceutical Affairs Law.

1. Patients taking four or more anti-hypertensive medications at Visit 1 2. Patients with known or suspected secondary hypertension (renovascular hypertension, primary aldosteronism, pheochromocytoma, etc.) 3. Patients whose mean seated DBP > 114 mmHg and/or mean seated SBP > 200 mmHg at Visit 1, Visit 2 or Visit 3 4. Patients with sustained ventricular tachycardia or other clinically relevant cardiac arrhythmias (AV-block II-III, atrial fibrillation etc.) 5. Patients with NYHA functional class heart failure III-IV 6. Patients with a history of myocardial infarction or cardiac surgery within last 6 3 months before signing the informed consent form 7. Patients with a history of coronary artery bypass surgery or percutaneous transluminal coronary angioplasty (PTCA) within last 3 months before signing the informed consent form 8. Patients with a history of unstable angina within last 3 months before signing the informed consent form 9. Patients with hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of aortic or mitral valve 10. Patients with a history of stroke or transient ischemic attack within last 6 months before signing the informed consent form 11. Patients with a history of sudden exacerbation of renal function with AT1 receptor antagonists or ACE inhibitors; post-renal transplant 12. Patients who have previously experienced characteristic symptoms of angioedema (such as facial, tongue, pharyngeal, or laryngeal swelling with dyspnea) during treatment with AT1 receptor antagonists or ACE inhibitors 13. Patients with known hypersensitivity to any component of the formulation, or a known hypersensitivity to sulfonamides or sulfonamide-derived drugs (e.g. thiazides) 14. Known, suspected or history of gout

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08

PRIMARY OUTCOMES:
Incidence of adverse events | 52 weeks
Changes in clinical laboratory tests (haematology, blood chemistry and urinalysis) | 52 weeks
Changes in electrocardiogram (ECG) | 52 weeks
Changes in blood pressure and pulse rate | 52 weeks

SECONDARY OUTCOMES:
Seated Diastolic Blood Pressure (DBP) control rate | after 12 and 52 weeks
Seated Systolic Blood Pressure (SBP) control rate | after 12 and 52 weeks
Seated DBP response rate | after 12 and 52 weeks
Seated SBP response rate | after 12 and 52 weeks
Seated blood pressure (BP) normality criteria | after 12 and 52 weeks
Changes in seated DBP | after 12 and 52 weeks
Changes in seated SBP | after 12 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Nippon Boehringer Ingelheim Co., Ltd.
Locations (3):
- Japan (3):
  - Boehringer Ingelheim Investigational Site, Hiroshima-shi, Hiroshima
  - Boehringer Ingelheim Investigational Site, Sapporo-shi, Hokkaido
  - Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/24834808